CLINICAL TRIAL: NCT00002261
Title: A Comparative Phase I Clinical Study of HIVAC-1e and Smallpox (Vaccinia) Vaccines in Previously (Vaccinia) Vaccinated and Unvaccinated Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Prevention
Other Study IDs: 063A; AI452-003001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; Smallpox Vaccine; HIV-1; AIDS Vaccines; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — Smallpox Vaccine; HIVAC-1e; VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: Smallpox Vaccine
Biological: HIVAC-1e
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To determine the physiological and immunological responses in healthy HIV seronegative adult volunteers vaccinated with a) the HIVAC-1e (vaccinia-HIV) vaccine expressing the envelope glycoproteins of HIV and b) the Wyeth smallpox vaccine. The parameters to be studied will include:

1. The course of physiological responses to vaccination, including (a) lesion development, progression, and resolution; (b) physiological changes such as temperature, malaise, itching at the site, etc. and (c) any observable AE.
2. The appearance, identity, quantity, and duration of humoral antibodies against HIV and vaccinia virus.
3. The appearance, identity, quantity, and duration of cell-mediated immunity against HIV and vaccinia virus.
4. The adequacy of a procedure using a special dressing to contain viral shedding from the vaccination site.
5. The safety, humoral and cellular immune responses of a booster injection of the recombinant subunit gp160 vaccine (MicroGeneSys) in HIVAC-1e recipients.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* All drugs, medications, and therapy which, by virtue of direct pharmacologic action or possible drug interaction, could influence the intended effects of the study vaccine or mask its side effects may be concomitantly administered only by prescription by the Principal Investigator and must be documented on the case report form (CRF).
* Any drug, even aspirin, which is administered after vaccination and during the follow up periods must be documented on the patient's CRF.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Failure to meet any criteria listed under Inclusion Criteria.
* Development of active eczema or other skin condition which would increase the risk of secondary vaccinia lesions.
* Appearance of serologic or clinical evidence of HIV infection prior to vaccination.
* Current evidence of clinically active viral infections such as Mononucleosis, Epstein-Barr Virus, or cytomegalovirus which may affect immunocompetence.
* Active and overt parasitic, mycobacterial, or pyogenic infections that affect tests designated in Inclusion Criteria.

Concurrent Medication:

Excluded:

* All drugs, medications and therapy not prescribed by the Principal Investigator, and not documented on the case report form (CRF).
* Any drug, even aspirin, which is administered after vaccination and during the follow up periods which is not documented on the patient's CRF.

Patients with the following are excluded:

* Failure to meet any criteria listed under Inclusion Criteria.
* Appearance of serologic or clinical evidence of HIV infection prior to vaccination.
* Current evidence of clinically active viral infections.
* Active and overt parasitic, mycobacterial, or pyogenic infections that affect tests designated in Inclusion Criteria.

Risk Behavior:

Patients who do not agree to behave sexually in a manner that will minimize the risk of HIV infection for the duration of the study are excluded.

Patients must:

* Be HIV seronegative.
* Have excellent general health.
* Be unable to bear children.
* Have no immediate household contacts, sex partners, intimate contacts.
* Be free of clinical skin diseases.
* Have signed an informed consent.
* Control subjects receiving Smallpox vaccine will also be selected under the same inclusion criteria. They may be recruited from low risk behavior populations; from laboratory and hospital employees providing service to the study who would normally require Smallpox vaccination; and may be heterosexual, homosexual, or bisexual.

Patients must agree to behave sexually in a manner that will minimize the risk of HIV infection for the duration of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol - Myers Squibb Co, Wallingford, Connecticut, United States